CLINICAL TRIAL: NCT04531397
Title: Efficacy and Safety of Dapagliflozin in Children With Proteinuric Chronic Kidney Disease : a Prospective, Randomized, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Dapagliflozin in Children With Proteinuric Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASOD.01
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Proteinuria; Chronic Kidney Diseases
Keywords: Angiotensin Converting Enzyme Inhibitors; Sodium-glucose co-transporter 2 inhibitors; Dapagliflozin
MeSH Terms: conditions — Proteinuria; Renal Insufficiency, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEI treatment (Placebo Comparator): Drug: ACEI will be given once daily
  Interventions: Drug: ACEI treatment
- Dapagliflozin+ACEI treatment (Experimental): Drug: ACEI, will be given once daily Drug: Dapagliflozin, will be given once daily
  Interventions: Drug: Dapagliflozin+ACEI treatment

INTERVENTIONS:
Drug: ACEI treatment — ACEI, will be given once daily based on body weight (0.2mg/kg/d-0.6mg/kg/d，max 20mg/d), for 24 weeks
  Other Names: Control group
  Arms: ACEI treatment
Drug: Dapagliflozin+ACEI treatment — Dapagliflozin will be given 10 mg/day (weight>30kg) or 5mg/day (weight≤30kg), for 24 weeks ACEI, will be given based on body weight (max 20mg/d), for 24 weeks.
  Other Names: Treatment group
  Arms: Dapagliflozin+ACEI treatment

SUMMARY:
We aim to investigate the antiproteinuric effect of adding Dapagliflozin to the standard of care in children with proteinuria.

DETAILED DESCRIPTION:
Blockers of renin angiotensin aldosterone system (RAAS) such as angiotensin converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARBs) are considered the standard of care in treatment of Proteinuric Chronic Kidney Disease. However, these agents lead to incomplete renal protection. The purpose of the study is to investigate the antiproteinuric effect of adding Dapagliflozin to the standard of care in children with proteinuria. In this study, participants were randomly assigned (1:1) to receive ACEI+Dapagliflozin (5mg or 10mg, based on body weight) or ACEI only once daily for 24 weeks. Prespecified outcomes includes changes in 24-hr proteinuria, albumin, eGFR (estimated glomerular filtration rate), blood pressure, body weight and so on.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to 18 years；
* Urinary protein excretion > 200 mg in a 24-hr urine collection；
* Without any immunosuppressant medications such as corticosteroids, CNIs and so on；
* Estimated GFR ≥ 60 ml/min/1.73m2（estimated with Schwartz formula）；
* No history of diabetes；
* On stable doses of ACE inhibitors or angiotensin receptor blockers (ARBs) for > 1 month；
* Willing to sign informed consent.

Exclusion Criteria:

* Autosomal dominant polycystic kidney disease or autosomal recessive polycystic kidney disease, lupus nephritis, or ANCA-associated vasculitis;
* Blood pressure less than 5th percentile of the same gender, age, and height;
* Uncontrolled urinary tract infection at screening;
* At risk for dehydration or volume depletion;
* Evidence of hepatic disease: an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) two times the upper limit of normal
* History of organ transplantation, cancer, liver disease;
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  1. History of active inflammatory bowel disease within the last six months;
  2. Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  3. Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months;
  4. Pancreatic injury or pancreatitis within the last six months;
* Participation in another therapeutic trial with an investigational drug within 30 days prior to informed consent;
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in 24 hour proteinuria | From baseline to week 12
  Urine will be collected for 24 hours and total urinary albumin excretion will be measured

SECONDARY OUTCOMES:
The change in 24 hour proteinuria | From baseline to week 24
  Urine will be collected for 24 hours and total urinary albumin excretion will be measured
The change in albumin from baseline to week 24 | Measured at baseline, weeks 4, weeks 8, weeks 12, weeks 24
  Serum albumin levels are repeated measurement data
The change in eGFR (estimated glomerular filtration rate) from baseline to week 24 | Measured at baseline, weeks 4, weeks 8, weeks 12, weeks 24
  eGFR will be evaluated using Schwartz formula (eGFR=k*height(cm)/serum creatinine(umol/L)), k=36.5), and eGFR are repeated measurement data
The change blood pressure from baseline to week 24 | Measured at baseline, weeks 4, weeks 8, weeks 12, weeks 24
  Blood pressure including systolic blood pressure (SBP) and diastolic blood pressure (DBP) are repeated measurement data
The change in body weight from baseline to week 24 | Measured at baseline, weeks 4, weeks 8, weeks 12, weeks 24
  Body weight are repeated measurement data and will be measured in the morning
The number of hypoglycemia episodes during the treatment | From baseline to week 24
  Patients will be asked to measure fasting blood glucose every morning and record the data by their parents during the treatment period. Hypoglycemia is defined as glucose level less than 3.9mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Shen, Profressor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No